CLINICAL TRIAL: NCT03914300
Title: Phase II Study of XL184 (Cabozantinib) in Combination With Nivolumab and Ipilimumab (CaboNivoIpi) in Patients With Radioiodine-Refractory Differentiated Thyroid Cancer Whose Cancer Progressed After One Prior VEGFR-Targeted Therapy
Brief Title: Testing the Combination of Cabozantinib, Nivolumab, and Ipilimumab (CaboNivoIpi) for Advanced Differentiated Thyroid Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-02220; NCI-2019-02220 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU-19088; 10240 (Other: Ohio State University Comprehensive Cancer Center LAO); 10240 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-06

CONDITIONS: Differentiated Thyroid Gland Carcinoma; Follicular Variant Thyroid Gland Papillary Carcinoma; Poorly Differentiated Thyroid Gland Carcinoma; Refractory Differentiated Thyroid Gland Carcinoma; Refractory Thyroid Gland Carcinoma; Tall Cell Variant Thyroid Gland Papillary Carcinoma; Thyroid Gland Follicular Carcinoma; Thyroid Gland Oncocytic Carcinoma; Thyroid Gland Papillary Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — Specimen Handling; cabozantinib; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cabozantinib S-malate, nivolumab, ipilimumab) (Experimental): Patients receive cabozantinib S-malate PO QD on days -14 to -1 prior to cycle 1, days 1-42 of cycles 1-4 and days 1-28 of subsequent cycles. Patients also receive nivolumab IV over 30 minutes on days 1, 15, and 29 of cycles 1-4 and day 1 of subsequent cycles and ipilimumab IV over 90 minutes on day 1 of cycles 1-4. Treatment repeats every 42 days for cycles 1-4 and every 28 days for subsequent cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI during screening, and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Cabozantinib S-malate; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL 184; XL-184; XL184
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase II trial studies how well cabozantinib, nivolumab, and ipilimumab work in treating patients with differentiated thyroid cancer that does not respond to radioactive iodine and that worsened after treatment with a drug targeting the vascular endothelial growth factor receptor (VEGFR), a protein needed to form blood vessels. Cabozantinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving cabozantinib, nivolumab and ipilimumab may work better than the usual approach consisting of chemotherapy with drugs such as doxorubicin, sorafenib, and lenvatinib for this type of thyroid cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the objective response rate, defined as the proportion of patients who have had a partial response (PR) or complete response (CR) within the first 6 months after initiation of therapy with cabozantinib S-malate (XL184 [cabozantinib]), nivolumab, and ipilimumab (CaboNivoIpi).

SECONDARY OBJECTIVES:

I. To assess duration of objective response (DOR), progression-free survival (PFS), and overall survival (OS).

II. To assess tolerability and adverse events of CaboNivoIpi in patients with differentiated thyroid cancer (DTC).

EXPLORATORY OBJECTIVES:

I. To correlate treatment response (Response Evaluation Criteria in Solid Tumors [RECIST] version [v]1.1) with tumor mutation status.

II. To correlate treatment response (RECIST v1.1) with frequency of tumor infiltrating lymphocytes in biopsies taken pre-treatment and after 12 weeks of CaboNivoIpi therapy.

III. To evaluate the effect of CaboNivoIpi on T cell receptor (TCR) repertoire and to identify the frequency of shared T cell clones between tumor and peripheral blood.

IV. To evaluate the effect of XL184 (cabozantinib) alone and of the CaboNivoIpi combination on peripheral blood mononuclear cells (PBMCs) and to correlate their frequency with treatment response (RECIST v1.1).

V. To evaluate the effect of XL184 (cabozantinib) alone and of the CaboNivoIpi combination on myeloid-derived suppressor cells (MDSCs) and to correlate their frequency with treatment response (RECIST v1.1).

VI. To correlate treatment response (RECIST v1.1) with programmed cell death protein 1 (PD-1) / programmed cell death-ligand 1 (PD-L1) expression in the primary/metastatic tumor.

OUTLINE:

Patients receive cabozantinib S-malate orally (PO) once daily (QD) on days -14 to -1 prior to cycle 1, days 1-42 of cycles 1-4 and days 1-28 of subsequent cycles. Patients also receive nivolumab intravenously (IV) over 30 minutes on days 1, 15, and 29 of cycles 1-4 and day 1 of subsequent cycles and ipilimumab IV over 90 minutes on day 1 of cycles 1-4. Treatment repeats every 42 days for cycles 1-4 and every 28 days for subsequent cycles in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) during screening, and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 6 weeks, and then every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed papillary thyroid cancer (PTC), follicular thyroid cancer (FTC), or Hurthle cell thyroid cancer (HTC). Follicular variant of PTC or any of the above mixed histology will be allowed, as well as tall cell, insular, or poorly-differentiated thyroid cancers. Patients with anaplastic thyroid cancers (ATC) or medullary thyroid cancers (MTC) are not eligible
* Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Patients must have radioactive iodine (RAI)-refractory/resistant disease as defined by one or more of the following criteria:

  * One or more measurable lesions that do not demonstrate RAI uptake,
  * Progressive disease (PD) (new lesion or progression of previously known lesions), as defined by RECIST v1.1, within 12 months of prior RAI therapy,
  * One or more measurable lesion present after cumulative RAI dose of > 600 mCi, or
  * Fluorodeoxyglucose (FDG)-positron emission tomography (PET) scan-positive disease (SUV >= 5 in tumor lesion)
* The patient's disease must have progressed on one line of VEGFR-targeted therapy (including, but not limited to, sorafenib, sunitinib, vandetanib, pazopanib, or lenvatinib, etc.) as defined by PD per RECIST v1.1 while receiving VEGFR-targeted therapy. Patients who have received more than one line of prior VEGFR-targeted therapy will not be eligible
* Prior external beam radiation to extra-osseous disease, systemic cytotoxic chemotherapy or BRAF- or non-VEGFR-targeted therapies will be allowed, provided that > 4 weeks has elapsed since receiving prior treatment. Radiation to bone metastases is allowed up to 2 weeks prior to initiation of study treatment
* Patients must be >= 18 years of age. Because no dosing or adverse event data are currently available on the use of XL184 (cabozantinib), nivolumab, or ipilimumab in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Patients must have recovered to baseline or =< Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grade 1 from toxicities related to any prior treatments, unless adverse event (AE)(s) are clinically nonsignificant and/or stable on supportive therapy
* Absolute neutrophils >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN); =< 3.0 x ULN for patients with Gilbert's syndrome
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional ULN
* Alkaline phosphatase =< 3.0 x institutional ULN; =< 5.0 x ULN with documented bone metastases
* Creatinine =< 1.5 x ULN OR creatinine clearance (CrCl) >= 50 mL/min (if using the Cockcroft-Gault formula)
* Serum albumin >= 2.8 g/dL
* Lipase < 2.0 x ULN and no radiologic or clinical evidence of pancreatitis
* Urine protein/creatinine ratio (UPCR) =< 1 mg/mg
* Serum phosphorus, calcium, magnesium, and potassium within institutional normal limits
* Prothrombin time (PT)/international normalized ratio (INR) and partial thromboplastin time (PTT) test < 1.3 x ULN
* Patients with a history of human immunodeficiency virus (HIV) infection must be on an effective anti-retroviral regimen utilizing agents that do not strongly induce or inhibit cytochrome P450 (CYP) 3A4, and must have an undetectable viral load measured within 6 months prior to study registration
* Patients with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. Patients with HCV infection who are currently on treatment are eligible if they have an undetectable HCV viral load
* The effects of XL184 (cabozantinib), nivolumab, and ipilimumab on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. WOCBP should use an adequate method to avoid pregnancy for 5 months after the last dose of study therapy. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity: 25 IU/L or equivalent units of human chorionic gonadotropin [hCG]) within 24 hours prior to the start of study therapy. Women must not be breastfeeding. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of < 1% per year. Men who receive study therapy and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of study therapy. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception
* WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level < 40 mIU/mL
* WOCBP and men who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 5 and 7 months, respectively, after the last dose of study therapy. These durations have been calculated using the upper limit of the half-life for nivolumab (25 days) and are based on the protocol requirement that WOCBP use contraception for 5 half-lives plus 30 days and men who are sexually active with WOCBP use contraception for 5 half-lives plus 90 days
* Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she (or the participating partner) must inform the treating physician immediately
* Patients must be able to swallow tablets
* Patients must be able to understand be willing to sign a written informed consent document
* Patients with impaired decision-making capacity (IDMC) will be eligible if they have a legally authorized representative (LAR) or caregiver available to assist them

Exclusion Criteria:

* Patients must not have had prior treatment with XL184 (cabozantinib), any MET-targeting tyrosine kinase inhibitor (TKI), or any MET-targeting monoclonal antibody (MetMAb), such as onartuzumab
* Patients must not have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T cell co-stimulation or immune checkpoint pathways
* Patients must not have a tumor invading or encasing any major blood vessels, and must not have evidence of tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum, or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of XL184 (cabozantinib)
* Patients must not have a diagnosis of another malignancy within 2 years before the first dose of study treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy. Adjuvant hormonal therapy for history of prostate or breast cancer is allowed
* Patients must not have received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies) within 4 weeks, or nitrosoureas/ mitomycin C within 6 weeks, before the first dose of study treatment. Patients may continue on bone-modifying agents (denosumab or bisphosphonates) with caution
* Patients must not have received radiation therapy:

  * To the thoracic cavity, abdomen, or pelvis within 4 weeks before the first dose of study treatment;
  * To bone metastases within 14 days before the first dose of study treatment;
  * To any other sites within 4 weeks before the first dose of study treatment
* Patients must not have clinically relevant, ongoing complications from prior radiation therapy. Palliative (limited-field) radiation therapy is permitted as long as the patient does not have disease progression according to RECIST v 1.1
* Patients must not have received any type of small molecule kinase inhibitor (including investigational kinase inhibitors) within 4 weeks before the first dose of study treatment
* Patients must not have received any other type of investigational agent within 4 weeks before the first dose of study treatment
* Patients must not have a corrected QT interval calculated by the Fridericia formula (QTcF) > 500 msec by electrocardiogram (EKG) within 28 days before the first dose of study treatment

  * Note: if a single EKG shows a QTcF with an absolute value > 500 msec, two additional EKGs at intervals of approximately 3 min must be performed within 30 min after the initial EKG, and the average of these three consecutive results for QTcF will be used to determine eligibility
* Patients should not have known, untreated brain metastases or leptomeningeal metastases because of poor prognosis and concerns that progressive neurologic dysfunction could confound the evaluation of neurologic and other adverse events. However, patients will be eligible if metastases have been treated, and there is no magnetic resonance imaging (MRI) evidence of progression for at least 4 weeks after treatment for metastases is complete and within 28 days prior to the first dose of study treatment
* Patients must not require concomitant treatment with oral anticoagulants (e.g., warfarin, direct thrombin, and factor Xa inhibitors) or platelet inhibitors (e.g., clopidogrel). The following anticoagulants are allowed:

  * Low-dose aspirin for cardioprotection (per local applicable guidelines),
  * Low-dose low molecular weight heparins (LMWH),
  * Therapeutic doses of LMWH are allowed in patients without known brain metastases who are on a stable dose of LMWH for at least 6 weeks before the first dose of study treatment, and who have had no clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor
* Patients must not require systemic corticosteroids treatment (>= 10 mg/day prednisone equivalents) or other immunosuppressive medications within 14 days prior to study drug administration. Inhaled or topical steroids and adrenal replacement doses < 10 mg/day prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if >= 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted, as is steroid pre-medication for contrast allergy
* Patients must not have a history of severe hypersensitivity reactions to any monoclonal antibodies
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study
* Patients must not require concomitant treatment with strong CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, or St. John's wort). Because lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list. Medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, patients will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients must not have uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association (NYHA) class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias
    * Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment within seven days prior to the first dose of study treatment
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or thromboembolic event (e.g., deep venous thrombosis [DVT], pulmonary embolism [PE]) within 6 months before first dose
  * GI disorders including those associated with a high risk of perforation or fistula formation:

    * The patient has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (e.g., Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction
    * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. Complete healing of an intra-abdominal abscess must be confirmed before first dose
  * Clinically significant hematuria, hematemesis, or hemoptysis or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose
  * Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation
  * Lesions invading or encasing any major blood vessels
  * Other clinically significant disorders that would preclude safe study participation

    * Serious non-healing wound/ulcer/bone fracture
    * Uncompensated/symptomatic hypothyroidism
    * Moderate to severe hepatic impairment (Child-Pugh B or C)
* Patients must not have had major surgery (e.g., GI surgery or removal or biopsy of brain metastasis) within 8 weeks before first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before the first dose of study treatment and from minor surgery (e.g., simple excision or tooth extraction) at least 10 days before the first dose. Patients with clinically relevant ongoing complications from prior surgery are not eligible
* Pregnant women are excluded from this study because XL184 (cabozantinib) has the potential for teratogenic or abortifacient effects, and the effects of nivolumab and ipilimumab on the developing fetus are not well known. Because there is an unknown but potential risk for AEs in nursing infants secondary to treatment of the mother, breastfeeding must be discontinued if the mother is treated with XL184 (cabozantinib), nivolumab, or ipilimumab
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including high dose systemic corticosteroids, should be excluded. These include but are not limited to: immune-related neurologic disease, such as multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, or myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, or autoimmune hepatitis. Patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patients with vitiligo, type I diabetes mellitus (DM), or endocrine deficiencies (e.g., thyroiditis) managed with replacement hormones, including physiologic corticosteroids, are eligible
* Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication, and patients with positive serology, (e.g., antinuclear antibodies [ANA] or anti-thyroid antibodies) should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2025-12-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bhavana Konda, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO
Locations (33):
- United States (33):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Konda B, Sherman EJ, Massarelli E, Nieva J, Muzaffar J, Morris JC 3rd, Ryder M, Ho AL, Agulnik M, Wei L, Handley D, Moses C, Jacob R, Wright J, Streicher H, Carson W, Shah MH. Cabozantinib Plus Ipilimumab/Nivolumab in Patients With Previously Treated Advanced Differentiated Thyroid Cancer. J Clin Endocrinol Metab. 2025 Feb 18;110(3):830-837. doi: 10.1210/clinem/dgae512. PMID 39133806

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Started | 11
Completed | 10
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 69 [44 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Defined as the proportion of patients who have had a partial response (PR) or complete response (CR) within the first 6 months after initiation of therapy.
Time Frame: Up to 6 months after initiation of therapy
Population: One participant was not evaluable for response as they experienced a grade 5 SAE before the first radiographic assesment
Measure: Number; unit: proportion of participants
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 10
proportion of participants | 0.1

2. Secondary Outcome: Treatment Related Adverse Events (TRAEs)
Description: Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. Frequency and severity of AEs and tolerability of the regimen will be collected and summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. Treatment related adverse events that occurred in >20% of participants are reported here.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 11
Participants
  Grade 1-2 TRAEs : Abdominal Pain | 3
  Grade 1-2 TRAEs : Alanine aminotransferase increased | 3
  Grade 1-2 TRAEs : Anemia | 3
  Grade 1-2 TRAEs : Anorexia | 4
  Grade 1-2 TRAEs : Aspartate aminotransferase increased | 5
  Grade 1-2 TRAEs : Diarrhea | 5
  Grade 1-2 TRAEs : Dysgeusia | 3
  Grade 1-2 TRAEs : Fatigue | 4
  Grade 1-2 TRAEs : Hypertension | 4
  Grade 1-2 TRAEs : Hypoalbuminemia | 3
  Grade 1-2 TRAEs : Hypokalemia | 4
  Grade 1-2 TRAEs : Muscle cramp | 3
  Grade 1-2 TRAEs : Nausea | 3
  Grade 1-2 TRAEs : Palmar-plantar erythrodysesthesia | 4
  Grade 1-2 TRAEs : Rash maculopapular | 5
  Grade 1-2 TRAEs : Weight loss | 4
  Grade 1-2 TRAEs : White blood cells decreased | 3
  Grade ≥ 3 TRAEs : Abdominal Pain | 0
  Grade ≥ 3 TRAEs : Alanine aminotransferase increased | 1
  Grade ≥ 3 TRAEs : Anemia | 0
  Grade ≥ 3 TRAEs : Anorexia | 0
  Grade ≥ 3 TRAEs : Aspartate aminotransferase increased | 1
  Grade ≥ 3 TRAEs : Diarrhea | 1
  Grade ≥ 3 TRAEs : Dysgeusia | 0
  Grade ≥ 3 TRAEs : Fatigue | 1
  Grade ≥ 3 TRAEs : Hypertension | 3
  Grade ≥ 3 TRAEs : Hypoalbuminemia | 0
  Grade ≥ 3 TRAEs : Hypokalemia | 0
  Grade ≥ 3 TRAEs : Muscle cramp | 0
  Grade ≥ 3 TRAEs : Nausea | 1
  Grade ≥ 3 TRAEs : Palmar-plantar erythrodysesthesia | 1
  Grade ≥ 3 TRAEs : Rash maculopapular | 0
  Grade ≥ 3 TRAEs : Weight loss | 0
  Grade ≥ 3 TRAEs : White blood cells decreased | 0

3. Secondary Outcome: Duration of Response
Description: From response (PR or CR) to documented progression
Time Frame: From response (PR or CR) to documented progression, assessed up to approximately 25 months
Population: One participant was not evaluable for response as they experienced a grade 5 SAE before the first radiographic assessment
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 10
months | 18.6 [11.8 to 25.4]

4. Secondary Outcome: Progression-free Survival
Description: Will be analyzed using Kaplan-Meier methods, resulting in median survival times with 95% confidence interval (CI).
Time Frame: From initiation of therapy to documented progression or death, whichever occurs first, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 11
months | 8 [3.0 to NA] — Upper threshold of confidence interval not met due to insufficient number of participants with events

5. Secondary Outcome: Overall Survival
Description: Will be analyzed using Kaplan-Meier methods, resulting in median survival times with 95% CI.
Time Frame: From initiation of therapy to death from any cause, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
Number analyzed (Participants) | 11
months | 19.2 [4.6 to NA] — Upper threshold of confidence interval not met due to insufficient number of participants with events

6. Other Pre Specified Outcome: Tumor Mutation Status
Description: Will be summarized using frequency and compared between responders and non-responders using chi-square test or Fisher's exact test, whichever is more appropriate.
Time Frame: Up to 2 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Tumor Infiltrating Lymphocyte in Biopsies
Description: Will be described graphically using boxplots or summary measures (e.g., mean and standard errors) at each time point. Will also explore how changes in these correlative markers may differ based on whether or not the patient achieved a response. To accomplish this, will utilize different plotting characters and colors for responses versus (vs.) not in the graphical analyses to help identify potential patterns, and summarize the changes quantitatively between responders and non-responders. Changes in levels will also be compared between responders and non-responders using two sample t-test or Wilcoxon test if the data is not normally distributed. Linear mixed effect models will also be used to examine the association of biomarkers over the time with the response. Potential confounders (patients' demographics and clinical characteristics) may also be included in the models.
Time Frame: Baseline up to 12 weeks after treatment start date
Reporting Status: Not Posted

8. Other Pre Specified Outcome: T Cell Receptor Repertoire in Peripheral Blood
Description: Will be described graphically using boxplots or summary measures (e.g., mean and standard errors) at each time point. Will also explore how changes in these correlative markers may differ based on whether or not the patient achieved a response. To accomplish this, will utilize different plotting characters and colors for responses vs. not in the graphical analyses to help identify potential patterns, and summarize the changes quantitatively between responders and non-responders. Changes in levels will also be compared between responders and non-responders using two sample t-test or Wilcoxon test if the data is not normally distributed. Linear mixed effect models will also be used to examine the association of biomarkers over the time with the response. Potential confounders (patients' demographics and clinical characteristics) may also be included in the models.
Time Frame: Baseline up to 12 weeks post treatment start date
Reporting Status: Not Posted

9. Other Pre Specified Outcome: T Cell Receptor Repertoire in Biopsies
Description: as for outcome 8
Time Frame: Baseline, 2 weeks after starting cabozantinib treatment, 12 weeks post treatment start date, and at the time of disease progression
Reporting Status: Not Posted

10. Other Pre Specified Outcome: PD-1/PD-L1 Expression in the Primary/Metastatic Tumor in Biopsies
Description: as for outcome 8
Time Frame: Baseline up to 12 weeks post treatment start date
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Peripheral Blood Mononuclear Cells
Description: as for outcome 8
Time Frame: as for outcome 9
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Circulating Myeloid-derived Suppressor Cells
Description: as for outcome 8
Time Frame: as for outcome 9
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab)
All-Cause Mortality (participants affected / at risk) | 7/11
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab) (N=11)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Alanine Aminotransferase increased (Investigations) | 1 (1)
Altered Mental Status (Nervous system disorders) | 1 (1)
Aspartate Aminotransferase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac troponin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Diastolic Heart Failure (Cardiac disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Gamma-Glutamyl Transferase (GGT) Increased (Investigations) | 1 (1)
Hepatitis (Infections and infestations) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Cabozantinib S-malate, Nivolumab, Ipilimumab) (N=11)
Abdominal pain (Gastrointestinal disorders) | 3 (7)
Adrenal insufficiency (Endocrine disorders) | 1 (37)
Alanine aminotransferase increased (Investigations) | 4 (25)
Alkaline phosphatase increased (Investigations) | 3 (27)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (12)
Anemia (Blood and lymphatic system disorders) | 5 (30)
Anorexia (Metabolism and nutrition disorders) | 5 (52)
Aspartate aminotransferase increased (Investigations) | 6 (39)
Axillary hydrandenitis suppurativa (Skin and subcutaneous tissue disorders) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (9)
Bloating (Gastrointestinal disorders) | 2 (4)
Blood bilirubin increased (Investigations) | 2 (3)
Blood lactate dehydrogenase increased (Investigations) | 4 (24)
Bruising (Injury, poisoning and procedural complications) | 2 (7)
Calcium decreased-intermittent (Metabolism and nutrition disorders) | 1 (5)
Chills (General disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 3 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Creatinine increased (Investigations) | 1 (3)
Depression (Psychiatric disorders) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 6 (54)
Dizziness (Nervous system disorders) | 1 (7)
Dry eye (Eye disorders) | 1 (4)
Dry mouth (Gastrointestinal disorders) | 1 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (5)
Dygeusia (Nervous system disorders) | 3 (21)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Ear pain (Ear and labyrinth disorders) | 1 (2)
Electocardiogram QT Corrected interval prolonged (Investigations) | 1 (4)
Fatigue (General disorders) | 6 (49)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (6)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (2)
General muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (10)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (10)
GGT increased (Investigations) | 3 (11)
Headache (Nervous system disorders) | 1 (13)
Hematuria (Renal and urinary disorders) | 1 (2)
Hemoptysis (Blood and lymphatic system disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Hidrandenitis suppurativa (Skin and subcutaneous tissue disorders) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (3)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 7 (40)
Hyperthyroidism (Endocrine disorders) | 1 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (23)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (18)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (18)
Hypokalemia (Metabolism and nutrition disorders) | 4 (12)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (19)
Hyponatremia (Metabolism and nutrition disorders) | 3 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (13)
Hpyophysitis (Endocrine disorders) | 1 (1)
Hypopituitarism (Endocrine disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (7)
Insomnia (Psychiatric disorders) | 1 (5)
Lipase increased (Investigations) | 2 (12)
Mean cell volume decreased (Investigations) | 1 (7)
Mucositis oral (Gastrointestinal disorders) | 3 (5)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 3 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Myocardial infarction (Cardiac disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (2)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (16)
Nasal pathway crustiness (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Nausea (Gastrointestinal disorders) | 5 (19)
Neuropathy (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (4)
Oral pain (Gastrointestinal disorders) | 1 (11)
Orthopnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain (General disorders) | 1 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (21)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 (31)
Paresthesia (Nervous system disorders) | 1 (2)
Platelet count decreased (Investigations) | 5 (11)
Platelet count increased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (6)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (44)
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (2)
Red blood cell count decreased (Investigations) | 1 (6)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Serum amylase increased (Investigations) | 1 (5)
Sinus pain (Nervous system disorders) | 4 (44)
Sinus tachycardia (Cardiac disorders) | 1 (5)
Skin rash, bilateral lower legs (Skin and subcutaneous tissue disorders) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (3)
Tail bone discomfort (Musculoskeletal and connective tissue disorders) | 1 (2)
Throat discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Thromboembolic event (Vascular disorders) | 1 (1)
Total protein decreased- intermittent (Investigations) | 1 (10)
Upper Respiratory Infection (Infections and infestations) | 1 (4)
Urinary tract infection (Infections and infestations) | 1 (4)
Vomiting (Gastrointestinal disorders) | 2 (8)
Weight loss (Investigations) | 6 (22)
White blood cell decreased (Investigations) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT03914300/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT03914300/ICF_001.pdf